CLINICAL TRIAL: NCT05379985
Title: A Multicenter Open-Label Study of RMC-6236 in Patients With Advanced Solid Tumors Harboring Specific Mutations in RAS
Brief Title: Study of RMC-6236 in Patients With Advanced Solid Tumors Harboring Specific Mutations in RAS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Revolution Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RMC-6236-001
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); Colorectal Cancer (CRC); Pancreatic Ductal Adenocarcinoma (PDAC); Advanced Solid Tumors
Keywords: KRAS; Non-small Cell Lung Cancer; Lung Cancer; Colorectal Cancer; Colon Cancer; Metastatic Cancer; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; NSCLC; CRC; PDAC; Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal; Colorectal Neoplasms; Colonic Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplastic Processes; Thoracic Neoplasms; Antineoplastic Agents; Melanoma; Gynecological Cancers; RAS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Lung Neoplasms; Colonic Neoplasms; Neoplasm Metastasis; Pancreatic Neoplasms; Carcinoma, Pancreatic Ductal; Intestinal Neoplasms; Gastrointestinal Neoplasms; Neoplastic Processes; Thoracic Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: RMC-6236 (Experimental): Enrollment into dose exploration may be from any advanced solid tumor type with KRAS p.G12 mutations.
  Enrollment into dose expansion/optimization may be from groups consisting of patients with a single histotype/genotype (for example, KRAS G12-mutated NSCLC, PDAC, CRC, RAS mutant NSCLC, Melanoma, gynecological cancer or other solid tumors not previously specified).
  RAS mutant is defined as any nonsynonymous mutation of KRAS, NRAS, or HRAS at codons 12, 13, or 61 (G12, G13, or Q61)
  Interventions: Drug: RMC-6236

INTERVENTIONS:
Drug: RMC-6236 — Oral Tablets

SUMMARY:
Evaluate the safety and tolerability of RMC-6236 in adults with specific RAS mutant advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/2, multicenter open-label study to evaluate the safety, tolerability, pharmacokinetics (PK), and clinical activity of escalating doses of RMC-6236 in adult patients with advanced solid tumors harboring specific RAS mutations, and to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose [RP2D] within investigated patient population groups. RMC-6236 is a potent, orally bioavailable RAS-MULTI(ON) inhibitor, selective for the active RAS(ON) form of both wild type and mutant variants of the canonical RAS isoforms (HRAS, NRAS, and KRAS).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor with specific KRAS G12 mutations (dose escalation) or RAS mutations (dose optimization/expansion) identified through deoxyribonucleic acid (DNA) sequencing. PDAC with wild-type RAS (expansion).
* Treatment naive or have received prior standard therapy appropriate for tumor type and stage
* Have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate organ function

Exclusion Criteria:

* Primary central nervous system (CNS) tumors
* Active, untreated brain metastases
* Known or suspected impairment of gastrointestinal function that may prohibit ability to swallow or absorb an oral medication
* History of any other unstable or clinically significant concurrent medical condition that would, in the opinion of the investigator, jeopardize the safety of a participant, impact their expected survival through the end of the study participation, and/or impact their ability to comply with the protocol prior/concomitant therapy

Other inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 754 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-07-26 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent Adverse Events (AEs) and serious AEs, including incidence and severity of findings in laboratory values and vital signs | up to 2.5 years
Number of Participants with Dose-Limiting Toxicity (DLT) | 21 days

SECONDARY OUTCOMES:
Maximum Observed Blood Concentration (Cmax) of RMC-6236 | up to 15 weeks
Time to Reach Maximum Blood Concentration (Tmax) of RMC-6236 | up to 15 weeks
Area Under Blood Concentration Time Curve (AUC) of RMC-6236 | up to 15 weeks
Elimination Half-Life of RMC-6236 (t1/2) | up to 15 weeks
Ratio of accumulation of RMC-6236 from a single dose to steady state with repeated dosing | up to 15 weeks
Overall Response Rate (ORR) | up to 2.5 years
  Overall response rate per RECIST v1.1
Duration of Response (DOR) | up to 2.5 years
  Duration of response per RECIST v1.1
Disease Control Rate (DCR) | up to 2.5 years
  Disease control rate per RECIST v1.1
Time to Response (TTR) | up to 2.5 years
  Time to response per RECIST v1.1
Progression-Free Survival (PFS) | up to 2.5 years
  Progression-free survival per RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Revolution Medicines, Inc., Study Director — Revolution Medicines, Inc.
Locations (16):
- United States (16):
  - UC Irvine/Chao Family Comprehensive Cancer Center, Orange, California
  - UCLA, Santa Monica, California
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas at Austin, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Next Oncology, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Next Oncology Virginia, Fairfax, Virginia

REFERENCES:
- [Derived] Jiang J, Jiang L, Maldonato BJ, Wang Y, Holderfield M, Aronchik I, Winters IP, Salman Z, Blaj C, Menard M, Brodbeck J, Chen Z, Wei X, Rosen MJ, Gindin Y, Lee BJ, Evans JW, Chang S, Wang Z, Seamon KJ, Parsons D, Cregg J, Marquez A, Tomlinson ACA, Yano JK, Knox JE, Quintana E, Aguirre AJ, Arbour KC, Reed A, Gustafson WC, Gill AL, Koltun ES, Wildes D, Smith JAM, Wang Z, Singh M. Translational and Therapeutic Evaluation of RAS-GTP Inhibition by RMC-6236 in RAS-Driven Cancers. Cancer Discov. 2024 Jun 3;14(6):994-1017. doi: 10.1158/2159-8290.CD-24-0027. Erratum In: Cancer Discov. 2025 Oct 6;15(10):2186. doi: 10.1158/2159-8290.CD-25-1519. PMID 38593348
- [Derived] Holderfield M, Lee BJ, Jiang J, Tomlinson A, Seamon KJ, Mira A, Patrucco E, Goodhart G, Dilly J, Gindin Y, Dinglasan N, Wang Y, Lai LP, Cai S, Jiang L, Nasholm N, Shifrin N, Blaj C, Shah H, Evans JW, Montazer N, Lai O, Shi J, Ahler E, Quintana E, Chang S, Salvador A, Marquez A, Cregg J, Liu Y, Milin A, Chen A, Ziv TB, Parsons D, Knox JE, Klomp JE, Roth J, Rees M, Ronan M, Cuevas-Navarro A, Hu F, Lito P, Santamaria D, Aguirre AJ, Waters AM, Der CJ, Ambrogio C, Wang Z, Gill AL, Koltun ES, Smith JAM, Wildes D, Singh M. Concurrent inhibition of oncogenic and wild-type RAS-GTP for cancer therapy. Nature. 2024 May;629(8013):919-926. doi: 10.1038/s41586-024-07205-6. Epub 2024 Apr 8. PMID 38589574
- [Derived] Schulze CJ, Seamon KJ, Zhao Y, Yang YC, Cregg J, Kim D, Tomlinson A, Choy TJ, Wang Z, Sang B, Pourfarjam Y, Lucas J, Cuevas-Navarro A, Ayala-Santos C, Vides A, Li C, Marquez A, Zhong M, Vemulapalli V, Weller C, Gould A, Whalen DM, Salvador A, Milin A, Saldajeno-Concar M, Dinglasan N, Chen A, Evans J, Knox JE, Koltun ES, Singh M, Nichols R, Wildes D, Gill AL, Smith JAM, Lito P. Chemical remodeling of a cellular chaperone to target the active state of mutant KRAS. Science. 2023 Aug 18;381(6659):794-799. doi: 10.1126/science.adg9652. Epub 2023 Aug 17. PMID 37590355